CLINICAL TRIAL: NCT06199739
Title: Safety of Immediate Weight-Bearing as Tolerated After Well-Reduced Geriatric Hip Fracture
Brief Title: Safety of Immediate Weight-Bearing as Tolerated After Well-Reduced Geriatric Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109046-E
Record Dates: First submitted 2023-07-07; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Bony Weight Bearing Disorder
Keywords: fracture reduction; proximal femur fracture; geriatrics
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early-Weight bearing (Experimental): Early Weight bearing was defined as starting Weight bearing within 48 h postoperatively, and WBAT referred to the adjustment of fracture site weight-bearing by pain tolerance.
  Interventions: Behavioral: Early-Weight bearing

INTERVENTIONS:
Behavioral: Early-Weight bearing — The patients began early weight bearing under attending physician and physiotherapist surveillance within 48 hours after surgery. Patients were instructed to stand up near the bed, and muscle power, gait stability, and pain tolerance were recorded. The physiotherapist instructed the patients to perform early mobilization and weight bearing as tolerable by self-adjustment of body weight distribution over the bilateral lower extremities, and walking assistance was used to prevent repeat falling accidents.

SUMMARY:
Purpose: Proximal femur fracture is a major traumatic injury in elderly populations; however, practical postoperative weight-bearing protocols are lacking. Therefore, the purpose of the present study was to investigate whether early weight-bearing status after proximal femur nail fixation is associated with any loss of reduction and evaluate the clinical outcomes of this intervention.

Patients and methods:

For this prospective single center clinical trial study, we recruited 14 proximal femur fracture cases, classified by AO/OTA 2018, receiving intramedullary nail fixation. Clinical outcomes included the Harris functional hip score and VAS pain score. Additionally, demographic data, radiological parameters, time to weight-bearing, mortality rate, medical and surgical complications, and final ambulation status were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AO/OTA type 31 fractures were included, and all fractures were classified using intraoperative fluoroscopy with traction on the fracture table.

Exclusion Criteria:

* Patients with pathological fractures, neurovascular insufficiency, ipsilateral lower extremity musculoskeletal injury, multiple fractures, or high risk of falling, including frequent falling accidents within 6 months, unsteady gait, ipsilateral neuropathy, limb weakness, and urinary incontinence were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 1 postoperatively
  The questionaire to patient. (HHS score 0-100,<60 poor,>80 good)
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 3 postoperatively
  The questionaire to patient(HHS score 0-100,<60 poor,>80 good)
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 6 postoperatively
  The questionaire to patient(HHS score 0-100,<60 poor,>80 good)
Harris Hip Functional score | Functional and radiographic evaluations was performed at months 12 postoperatively
  The questionaire to patient(HHS score 0-100,<60 poor,>80 good)

SECONDARY OUTCOMES:
visual analog pain score | Record at months 1 postoperatively
  Independent assessor (VAS:0-10)
visual analog pain score | Record at months 3 postoperatively
  Independent assessor(VAS:0-10)
visual analog pain score | Record at months 6 postoperatively
  Independent assessor(VAS:0-10)
visual analog pain score | Record at months 12 postoperatively
  Independent assessor(VAS:0-10)
Complication | Functional and radiographic evaluations were performed at months 1, 3, 6, and 12 postoperatively
  Loss of reduction, malunion or nonunion

CONTACTS AND LOCATIONS:
Locations (1):
- Far-Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided